CLINICAL TRIAL: NCT07364747
Title: Protective Effect of Acetylcysteine Against Cisplatinum-Induced Ototoxicity: A Randomized Controlled Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naphassakorn Opasatian, Protective Effect of Acetylcysteine against Cisplatinum-Induced Ototoxicity: A Randomized Controlled Trial, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COA no. SI 655/2024
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cisplatin-induced Ototoxicity; Sensorineural Hearing Loss; Ototoxicity; Ototoxicity, Drug-Induced
Keywords: Cisplatin-induced Ototoxicity; Sensorineural Hearing Loss; Ototoxicity
MeSH Terms: conditions — Hearing Loss, Sensorineural; Ototoxicity | interventions — Acetylcysteine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N acetylcysteine (Experimental): NAC at a dosage of 150 mg/kg in 5%DW 200 mL intravenous 4-6 hour after completion of cisplatin
  Interventions: Drug: Acetyl cysteine
- Control Group (Placebo Comparator): Normal saline 200 mL intravenous 4-6 hour after completion of cisplatin
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Acetyl cysteine — N-acetylcysteine at a dosage of 150 mg/kg in 5%DW 200 mL intravenous 4-6 hour after completion of cisplatin which dosage more than 50 mg/m2 and planned cumulative dose more than 200 mg/m2
  Arms: N acetylcysteine
Drug: Normal Saline — Normal saline 200 mL intravenous 4-6 hour after completion of cisplatin which dosage more than 50 mg/m2 and planned cumulative dose more than 200 mg/m2
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of N-acetylcysteine (NAC) in preventing cisplatin-induced ototoxicity in patients receiving cisplatin-based chemotherapy. Cisplatin is a highly effective chemotherapeutic agent but often leads to permanent hearing loss (ototoxicity) as a significant side effect. This study investigates whether the administration of NAC as an otoprotective agent can reduce or prevent the decline in hearing sensitivity, particularly at extended high frequencies, as measured by audiometry and distortion product otoacoustic emissions (DPOAE).

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, controlled] trial to investigate the protective effects of N-acetylcysteine (NAC) against cisplatin-induced hearing loss.

Patients scheduled to receive cisplatin chemotherapy will be enrolled. The primary objective is to compare the changes in hearing thresholds between the intervention group (receiving NAC) and the control group. Hearing function will be comprehensively evaluated using:

Pure-tone Audiometry (including Extended High-Frequency Audiometry).

Distortion Product Otoacoustic Emissions (DPOAE) to assess outer hair cell function.

Evaluations will be conducted at baseline (before chemotherapy) and before every cycle of cisplatin administration and 1 month and 4 month after completion . Statistical analysis will include descriptive statistics and comparative tests (such as Unpaired T-tests or Generalized Estimating Equations) to determine the significance of hearing threshold shifts. The study aims to provide evidence on the feasibility and effectiveness of NAC in preserving auditory function in cancer patients.

Outcome Measures

Primary Outcome Measure:

- Compare hearing levels between the N-Acetylcysteine group and the placebo group in patients receiving cisplatin, at one month after the completion of treatment by audiometry in term of each frequency and Pure tone average of 500,1000,2000 and 500,1000,2000,4000 and DPOAE

Secondary Outcome Measure:

* Compare hearing levels between the N-Acetylcysteine group and the placebo group in patients receiving cisplatin, prior to each cisplatin cycle administration and 4 months after completion of treatment by audiometry in term of each frequency and Pure tone average of 500,1000,2000 and 500,1000,2000,4000 and DPOAE
* The subsequent otologic symptoms following cisplatin therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* Patients scheduled to receive high-dose cisplatin-based chemotherapy regimens with a projected cumulative cisplatin dose of > 200 mg/m2 and each dose > 50 mg/m2
* Patients may receive concurrent chemotherapy with non-ototoxic agents
* Patients may receive concurrent radiation therapy to the skull base, provided the radiation dose does not exceed the toxic threshold for ototoxicity
* Patients receiving an appropriate antiemetic regimen consisting of Olanzapine or Neurokinin-1 (NK1) receptor antagonists
* Patients receiving medical treatment at Siriraj Hospital.

Exclusion Criteria:

* Patients diagnosed with Nasopharyngeal Carcinoma (CA nasopharynx).
* Patients with a history of head and neck radiation therapy where the radiation dose to the cochlea exceeded 9 Gy or the dose to the eustachian tube exceeded 50 Gy on both sides.
* Patients who have received N-acetylcysteine (NAC) within 2 weeks prior to the start of the study.
* Patients who have received other ototoxic drugs within 2 weeks prior to or during the study, including but not limited to:

Aminoglycoside antibiotics, Vancomycin, Loop diuretics (e.g., Furosemide), High-dose Aspirin, Antimalarial drugs (e.g., Quinine)

- Patient with a known allergy or hypersensitivity to acetylcysteine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
- Extended high frequency audiogram - DPOAE | 1 month after completion of cisplatin therapy
  Compare hearing levels between the N-Acetylcysteine group and the placebo group in patients receiving cisplatin, at one month after the completion of treatment by audiometry in term of each frequency and Pure tone average of 500,1000,2000 and 500,1000,2000,4000 and DPOAE

SECONDARY OUTCOMES:
- Extended high frequency audiogram - DPOAE | Prior to each cisplatin cycle administration and 4 months after completion of treatment
  - Compare hearing levels between the N-Acetylcysteine group and the placebo group in patients receiving cisplatin, prior to each cisplatin cycle administration and 4 months after completion of treatment by audiometry in term of each frequency and Pure tone average of 500,1000,2000 and 500,1000,2000,4000 and DPOAE
The subsequent otologic symptoms following cisplatin therapy | 1 month and 4 month after treatment
  The subsequent otologic symptoms following cisplatin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kanthong Thongyai, Master, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkoknoi, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to ensure the protection of participant privacy and to comply with the current institutional ethics committee guidelines